CLINICAL TRIAL: NCT04079374
Title: Open, Randomized, Comparative, Multicenter Study in Parallel Groups of the Efficacy, Safety, Immunogenicity of Etanercept and Enbrel, Lyophilisates for Solution for Subcutaneous Injection, in Patients With Rheumatoid Arthritis
Brief Title: Comparative Efficacy, Safety and Immunogenicity Study of Etanercept and Enbrel
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Joint Stock Company "Farmak" (Industry)
Collaborators: Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FM-ENRT-17
Record Dates: First submitted 2019-09-03; First posted 2019-09-06 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Rheumatoid Arthritis
Keywords: Etanercept; Enbrel
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Etanercept (Experimental): Patients receive Etanercept in the form of subcutaneous injections at a dose of 25 mg 2 times a week for 24 weeks.
  Interventions: Drug: Etanercept
- Enbrel (Active Comparator): Patients receive Enbrel in the form of subcutaneous injections at a dose of 25 mg 2 times a week for 24 weeks.
  Interventions: Drug: Enbrel

INTERVENTIONS:
Drug: Etanercept — Subcutaneous injections
  Other Names: L04AB01
  Arms: Etanercept
Drug: Enbrel — Subcutaneous injections
  Other Names: L04AB01; etanercept
  Arms: Enbrel

SUMMARY:
The Study objectives are:

1. To compare the efficacy and safety of Etanercept, lyophilisate for solution for injection and Enbrel, lyophilisate for solution for subcutaneous injection, which are used as subcutaneous injections at a dose of 25 mg 2 times a week for 24 weeks in combination with methotrexate in patients with rheumatoid arthritis.
2. To prove the therapeutic equivalence of Etanercept, lyophilisate for solution for injection and Enbrel, lyophilisate for solution for subcutaneous injection in patients with rheumatoid arthritis.
3. To evaluate the immunogenicity of Etanercept, lyophilisate for solution for injection.

DETAILED DESCRIPTION:
This is an open-label, randomized, comparative, multicentre study in parallel groups of the efficacy, safety and immunogenicity of Etanercept, lyophilisate for solution for injection and Enbrel, lyophilisate for solution for subcutaneous injection, in patients with rheumatoid arthritis.

Total duration of patient participation in the study will be 49-52 weeks. Of these: screening - up to 4 weeks, treatment - 24 weeks, follow-up after treatment - 4 weeks, evaluation of the study drug immunogenicity - 52 weeks after the treatment initiation.

Patients receive Etanercept or Enbrel (depending on the group) in the form of subcutaneous injections at a dose of 25 mg 2 times a week for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* patients of both sexes, from 18 to 75 years old;
* body weight > 45 kg;
* patients diagnosed with: rheumatoid arthritis (RA) of moderate and high activity, according to the classification of RA criteria of the American College of Rheumatology (ACR) and the European League Against Rheumatism (EULAR) of 2010;
* functional class I, II or III according to the Classification of the Functional Class of the RA of the American College of Rheumatology (ACR);
* number of painful joints (NPJ) ≥ 6 (68 joints examined), number of swollen joints (NSJ) ≥6 (66 joints examined);
* ESR (Erythrocyte sedimentation rate)≥ 28 mm/hour or СRP (C - reactive protein) > 7.0 mg/dl;
* patient who receive methotrexate for at least 12 weeks at doses of 7.5-20 mg/week (orally or parenterally), and the dose and route of administration of methotrexate was not changed for 4 weeks before randomization;
* patient who stopped therapy with other basic antirheumatic drugs, except methotrexate, and completed the wash-out period for these drugs of at least five half-life periods, but not less than 2 weeks (whichever is longer);
* if a patient takes NSAIDs (Nonsteroidal anti-inflammatory drugs), the dose of the drug should be stable within 2 weeks before randomization;
* if a patient takes oral glucocorticosteroids, the dose should be ≤10 mg/day of prednisolone (or equivalent) and be stable for 2 weeks before randomization;
* women of childbearing age and men who have partners, who have agreed to use reliable contraceptive methods during the entire study period and within 3 months after its termination. Reliable methods of contraception include: intrauterine devices, double-barrier method or state after surgical sterilization and vasectomy;
* signed informed consent of participants to participate in this study, which was obtained before any screening procedures, including discontinuation of forbidden-drugs.

Exclusion Criteria:

* known hypersensitivity to Etanercept or other components of the study drugs;
* other rheumatic diseases, autoimmune diseases, connective tissue diseases, immunodeficiency (e.g. psoriasis, psoriatic arthritis, primary Sjogren syndrome, systemic lupus erythematosus or demyelinating diseases such as multiple sclerosis);
* septic arthritis within 12 months before screening; purulent arthritis of prosthetic joints;
* acute or frequent recurrent chronic, local or generalized infections (bacterial/fungal/viral) or sepsis, or history of recurrent infections, or increased risk of developing infections or sepsis;
* an active form of tuberculosis; the history of the ineffective treatment of tuberculosis; latent tuberculosis or risk of developing tuberculosis (e.g., contact with patients who have an active form of tuberculosis, shortly before screening);
* severe interstitial lung diseases (bronchial asthma, chronic obstructive pulmonary disease, bronchiectasis, fibrosis);
* malignant diseases, including history (except successfully treated non-metastatic basal cell or squamous cell skin cancer or cervical cancer);
* congestive heart failure of class III or IV, according to New York Heart Association criteria, or unstable angina;
* uncontrolled diabetes mellitus, uncontrolled arterial hypertension;
* abnormal laboratory parameters at screening:
* haemoglobin < 100.0 g/L;
* platelets < 125 *10^9 cell/L;
* leukocytes < 3.5 *10^9 cell/L,
* absolute neutrophil count < 1.5 *10^9 cell/L;
* absolute lymphocyte count < 0.8 *10^9 cell/L;
* ASТ (Aspartate aminotransferase), АLТ (Alanine aminotransferase) 3 and more times higher than the upper limit of normal and serum total bilirubin 2 and more times higher than the upper limit of normal;
* serum creatinine 2 times or higher than the upper limit of normal;
* history of clinically significant or uncontrolled diseases of the respiratory system, liver, kidney, blood, gastrointestinal tract, endocrine system, immune system, skin, nervous system (including demyelinating disorders), cardiovascular system, or history of an autoimmune or mental disorder, or any condition which, in the opinion of the Investigator, can pose a threat to the safety of a patient, affect the study results or prevent a patient from completing the study;
* hepatitis В, С;
* scheduled surgical intervention including joint replacement during the study;
* recent chickenpox;
* oral and gastrointestinal ulcers;
* pregnancy, breastfeeding;
* history of alcohol or drug abuse;
* vaccination with live or attenuated vaccines within 4 weeks before the screening, or scheduled vaccination during the study, or within 3 months after the last dose of the study/reference drug;
* previous treatment with any other GEBD (genetically engineered biological drugs) (GEBD) for rheumatoid arthritis (including, tocilizumab, adalimumab, anakinra, abatacept, infliximab, rituximab, golimumab, Etanercept, certolizumab) or tofacitinib;
* use of systemic or intraarticular corticosteroids, except prednisolone at a dose of≤10 mg/day orally, or equivalent to GCS (Glucocorticosteroids) within 2 weeks before randomization;
* use of alkylating agents (e.g. cyclophosphamide, chlorambucil) within 6 months before randomization;
* use of intravenous or oral antimicrobial agents 4 weeks before randomization; simultaneous participation in any other clinical study, or participation in a clinical study within 3 months before screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2018-09-03 (Actual); Primary Completion 2021-12-03 (Estimated); Study Completion 2023-12-03 (Estimated)

PRIMARY OUTCOMES:
Number of patients with ACR20 (American College of Rheumatology 20 criteria) response | at 24 week of treatment.
  ACR20 responders are subjects with at least 20% improvement from Baseline for tender joint count (TJC), swollen joint count (SJC), and at least 3 of the 5 remaining core set measures:
  1. Health Assessment Questionnaire-Disability Index (HAQ-DI),
  2. C-reactive Protein (CRP),
  3. Patient's Assessment of Arthritis Pain-Visual Analog Scale (PAAP-VAS),
  4. Patient's Global Assessment of Disease Activity-Visual Analog Scale (PtGADA-VAS),
  5. Physician's Global Assessment of Disease Activity-Visual Analog Scale (PhGA-VAS)

SECONDARY OUTCOMES:
Number of patients with ACR50 (American College of Rheumatology 50 criteria) response | at 4, 8 and 12 weeks of treatment
  ACR50 responders are subjects with at least 50% improvement from Baseline for tender joint count (TJC), swollen joint count (SJC), and at least 3 of the 5 remaining core set measures:
  1. Health Assessment Questionnaire-Disability Index (HAQ-DI),
  2. C-reactive Protein (CRP),
  3. Patient's Assessment of Arthritis Pain-Visual Analog Scale (PAAP-VAS),
  4. Patient's Global Assessment of Disease Activity-Visual Analog Scale (PtGADA-VAS),
  5. Physician's Global Assessment of Disease Activity-Visual Analog Scale (PhGA-VAS)
Number of patients with ACR70 (American College of Rheumatology 70 criteria) | at 4, 8 and 12 weeks of treatment
  ACR70 responders are subjects with at least 70% improvement from Baseline for tender joint count (TJC), swollen joint count (SJC), and at least 3 of the 5 remaining core set measures:
  1. Health Assessment Questionnaire-Disability Index (HAQ-DI),
  2. C-reactive Protein (CRP),
  3. Patient's Assessment of Arthritis Pain-Visual Analog Scale (PAAP-VAS),
  4. Patient's Global Assessment of Disease Activity-Visual Analog Scale (PtGADA-VAS),
  5. Physician's Global Assessment of Disease Activity-Visual Analog Scale (PhGA-VAS)
Number of patients who achieved remission (DAS28(Disease Activity Score 28)<2.6) and low disease activity (DAS28≤3.2) | at 12 and 24 weeks of treatment
  The DAS28 is a combined index for measuring disease activity in RA. The index includes swollen (range 0-28) and tender (range 0-28) joint counts, acute phase response (ESR in mm/hr), and general health status (participant global assessment of disease activity using VAS, range 1-100 mm).
  DAS28, which uses a 28-joint count, is derived from the original DAS, which includes a 44-swollen joint count.
  The DAS28 scale ranges from 0 to 10, where higher scores indicate worsening. DAS28 <2.6 equals (=) remission
Changes in activity index DAS28 | at 4, 8, 12 and 24 weeks of treatment
  Changes in activity index compared to baseline. The DAS28 index takes into account information on safety and swelling of 28 joints, ESR and patients' global health assessment according to VAS.
  Calculate DAS28 from the expression:
  DAS28 = 0.56√NPJ + 0.28√NSJ + 70lnESR + 0.014PGAH, where NPJ - number of painful joints at palpation (28 examined), NSJ - number of swollen joints (28 examined), PGAH - patient's global assessment of health in millimetres in 100 mm Visual Analog Scale (VAS), ESR - rate of erythrocyte sedimentation in mm/h, ln - natural logarithm.
  According to the ACR criteria, the levels of the disease activity depending on the values of DAS28, are ranked as:
  remission - DAS28 <2.6; low - DAS28 ≤3.2; moderate - DAS28 3.3-5.1; high - DAS28 >5.1.
  To calculate DAS28, use the official online calculator: http://www.das-score.nl/das28/DAScalculators/dasculators.html and https://www.das-score.nl/das28/DAScalculators/dasculators.html
Changes in functional state of patients according to questionnaire HAQ -(Health Assessment Questionnaire- data) | at 4, 8, 12 and 24 weeks of treatment compared to baseline.
  Changes in functional state of patients according to questionnaire HAQ DI -(Health Assessment Questionnaire Disability Index) compared to baseline. It includes the categories of dressing and grooming, arising, eating, walking, hygiene, reach, grip and common daily activities. It asks patients about the amount of difficulty they experience in these activities as well as the use of aids and/or devices. The HAQ has a numeric rating scale (NRS) (13) to assess pain on a scale from 0 to 10.Grades to evaluate the treatment efficacy using the HAQ DI. The minimal clinically significant change in the HAQ DI, which corresponds to the difference in parameters before and after treatment, is equal to 0.22. НАQ < 0.22 points - no effect; 0.22 ≤ ∆ НАQ ≤ 0.36 - lowest effect (20% improvement according to ACR criterion); 0.36 ≤ ∆ HAQ < 0.80 - satisfactory effect (50% improvement according to ACR criterion); HAQ ≥ 0.80 points - highest effect (70% improvement according to ACR criterion).

CONTACTS AND LOCATIONS:
Overall Officials: Mykola Stanislavchuk, MD, PhD, Principal Investigator — Vinnitsa Regional Clinical Hospital Named after N.I.Pirogov
Locations (10):
- Ukraine (10):
  - PU Kryvyi Rih City Clinical Hospital №2 of the Dnipropetrovsk regional council, Kryvyi Rih, Dnipropetrovsk Oblast
  - PU Kryvyi Rih City Clinical Hospital №8 of the Dnipropetrovsk regional council, Kryvyi Rih, Dnipropetrovsk Oblast
  - Ivano-Frankivsk Central City Clinical Hospital, Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Communal non-commercial enterprise of Kharkiv Regional Council Regional Hospital of the war veterans, Kharkiv, Kharkivs’ka Oblast’
  - Municipal nonprofit enterprise City Multidisciplinary Hospital № 18 of Kharkiv City Council, Kharkiv, Kharkivs’ka Oblast’
  - Khmelnytskyi Regional Hospital, Khmelnytskyi, Khmelnytskyi Oblast
  - Communal noncommercial enterprise of Lviv Regional Council Lviv Regional Clinical Hospital, Lviv, Lviv Oblast
  - Ternopil University Hospital, Ternopil, Ternopil Oblast
  - Vinnitsa Regional Clinical Hospital Named After N.I.Pirogov, Vinnitsa, Vinnitsa Region
  - Municipal Institution O.Herbachevskiy Regional State Clinical Hospital, Zhytomyr, Zhytomyr Oblast